CLINICAL TRIAL: NCT06838715
Title: Role of Steroids and Extended Scorpion Anti-Venom Use in Cardiac Affection Among Scorpion Stung Pediatric Cases
Acronym: Scorpion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yousef Ahmed Yousef Hasan, Lecturer of Pediatrics, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Scorpion in Pediatrics
Record Dates: First submitted 2024-12-16; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-09

CONDITIONS: Scorpion Envenomation
MeSH Terms: conditions — Scorpion Stings | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group of non extended anti-venom: (Active Comparator): About 20 Patients treated with classical non extended anti-venom regimen as 3-5 ampoules by injection and supportive measure only with evaluation of cytokine 6 hours, 24 hours and 72 hours or relief of symptoms after the sting.
  Interventions: Drug: Dexamethasone
- Group of Dexamethazone (Active Comparator): About 20 Patients treated with Dexamethazone (The dose as: 0.2 mg/kg/day in week1, 0.15 mg/kg/day in week 2, 0.075 mg/kg/day in week) besides supportive measures with evaluation of cytokine 6 hours, 24 hours and 72 hours or relief of symptoms after the sting.
  Interventions: Drug: Dexamethasone
- Group of extended antivenom regimen (Active Comparator): About 20 Patients treated with extended antivenom regimen as 3-5 ampoules by injection besides supportive measures with evaluation of cytokine 6 hours, 24 hours and 72 hours or relief of symptoms after the sting.
  Interventions: Drug: Dexamethasone
- Group of Dexamethazone and extended antivenom regimen (Active Comparator): About 20 Patients treated with Dexamethazone (The dose as: 0.2 mg/kg/day in week1, 0.15 mg/kg/day in week 2, 0.075 mg/kg/day in week) and extended antivenom regimen as 3-5 ampoules by injection besides supportive measures with evaluation of cytokine evaluation of cytokine 6 hours, 24 hours and 72 hours or relief of symptoms after the sting.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Assessing the relation between the level of cytokines (interleukins and tumor necrosis factor alpha) and the development of cardiac complications associated with scorpion envenomation among pediatric patients. and Evaluating the role of the use of Dexamethasone and/or extended anti-venom administration on cardiac function and outcome in pediatric cases.
  Other Names: Scorpion Anti Venom

SUMMARY:
Scorpion envenomation is considered a serious public health issue in the Middle East and Northern Sahara . According to the world health organization (WHO), around 1.2 to 1.5 million individuals are suspected to scorpion stings annually in Middle East; with 3000 to 5000 deaths rate .

DETAILED DESCRIPTION:
In Egypt, the percent of scorpion cases was 1.6% of all patients presented to Ain Shams University Poison Control Center during 2019.Initially within 1-2 hours of sting hypotension and bradycardia are encountered followed by hypotension and tachycardia between 4 and 48 hours due to severe left ventricular dysfunction and hypotension alone with good volume pulse and warm extremities is observed later in the recovery stage.

Cardiopulmonary problems such pulmonary edema and/or cardiogenic shock are the key characteristics of severe cases.Myocardial ischemia, release of catechol amines, and the direct impact of scorpion venom on cardiac fibers are the main three explanations to these cardiac complications.

Inflammation is one of the key processes involved in the pathogenesis. Neurotoxins can cause the release of inflammatory mediators. Increased pulmonary vascular permeability following the release of inflammatory mediators, such as platelet activating factor, leukotrienes, and prostaglandins had been suggested to explain the development of cardiogenic pulmonary edema.

Troponin is the biomarker of choice for the detection of cardiac injury. Cardiac troponin I (cTnI) isoform is predominant in myocardial tissue .Increased serum levels of pro-inflammatory cytokines, interleukins and tumor necrosis factor alpha had also been observed in many experimental studies following scorpion envenomation in plasma and in rat lungs respectively and on humans.

Scorpion Anti-Venom has a significant role in life saving of stung patients, but there is still a conflict about the duration of its administration mainly after occurrence of myocardial toxicity in stung patients. Corticosteroids are known to decrease the level of inflammatory mediators produced during the process of inflammation including cytokines. Dexamethasone is steroid with powerful anti-inflammatory effect that works by calming down body's immune response to reduce pain, itching and swelling .

ELIGIBILITY:
Inclusion Criteria:

- Patients with scorpion stings and diagnosed as grade 1, 2 & 3 (according to recent history of scorpion sting and clinical presentation at the time of admission) .

Exclusion Criteria:

* Patients with history of cardiac disease, OR previous cardiac operation and or previous abnormal cardiac investigations .
* Patients with history of chronic renal, hepatic, chest or CNS diseases .
* Patients with chronic inflammatory diseases such as auto-immune diseases, with chronic use of corticosteroids .
* Envenomated cases that are described as grade 4 scorpion envenomation.
* Cases of scorpion sting above age of 18 years.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of steroids and anti-venom regimen | 7 days
  80 of patients will take Treatment of the scorpion sting by using steroids and extended anti-venom regimen and assessing them after the treatment to see if they in need of intubation or ICU admission or hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Khalifa Mohamed, lecturer, Study Director — Assiut University; Nagwa Mahmoud Ali, professor, Study Chair — Assiut University; Hala Mohamed Fathi, professor, Study Chair — Assiut University
Locations (1):
- Assiut University Pediatric Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abroug F, Ouanes-Besbes L, Tilouche N, Elatrous S. Scorpion envenomation: state of the art. Intensive Care Med. 2020 Mar;46(3):401-410. doi: 10.1007/s00134-020-05924-8. Epub 2020 Mar 3. PMID 32125457